CLINICAL TRIAL: NCT00006512
Title: Characterizing a 5P-Linked BHR Susceptibility Locus
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 948; R01HL066533 (NIH)
Record Dates: First submitted 2000-11-20; First posted 2000-11-21 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

SUMMARY:
To identify the predisposing genes responsible for asthma and bronchial hyperresponsiveness (BHR) at region 5p13.3 in an inbred Hutterite community.

DETAILED DESCRIPTION:
BACKGROUND:

Asthma is the most common chronic disease in industrialized nations, affecting more than10 million people in the U.S. alone. Familial aggregation and concordance rates in monozygotic twins have suggested a genetic component to asthma. Dr. Ober and colleagues have been conducting studies on the genetics of asthma and atopy in the Hutterites, an inbred population of European origins that practices a communal lifestyle. A genome-wide screen with 564 markers (average spacing 6 cM) was completed in an extended pedigree of 717 Hutterites who were well characterized with respect to asthma, atopy, and related phenotypes. These individuals are descendants of only 64 ancestors who lived in the early 1700's to the early 1800's. Evidence for linkage with bronchial hyperresponsiveness (BHR) by the likelihood ratio test extended over 30 centimorgans (cM) on chromosome 5p, with P-values as small as 0.001. Additional evidence for linkage at this same location was evident by the transmission disequilibrium test (P=0.0061). Typing additional markers in this region identified a critical region of 2.4 cM, corresponding to 1.5 Mb of DNA, and a high risk haplotype that is over transmitted to affected individuals.

The study was conducted in response to a Request for Applications, "Positional Candidate Approaches in Asthma Gene Discovery" released in Ocatober, 1999.

DESIGN NARRATIVE:

Dr. Ober and colleagues characterized the 5p-linked BHR susceptibility locus in the inbred Hutterites by positional cloning and replicating these findings in outbred, ethnically diverse populations. They examined single nucleotide polymorphisms (SNPs) spaced about 10 kb apart in each gene, and assessed the evidence for over transmission to affected offspring with each SNP and SNP haplotypes. Associations in the Hutterites were replicated in two outbred samples (a Caucasian sample from Germany, and an African American sample from Chicago). The functional effects of associated variants were assessed by in vitro assays as well as by genotype-phenotype studies in outbred samples that had been evaluated for asthma and atopy phenotypes. Identifying asthma or BHR susceptibility loci may identify novel pathways in asthma pathogenesis, thereby allowing for the development of new therapies and intervention strategies for these common diseases.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-09; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carole Ober — University of Chicago

REFERENCES:
- [Background] Ober C. Susceptibility genes in asthma and allergy. Curr Allergy Asthma Rep. 2001 Mar;1(2):174-9. doi: 10.1007/s11882-001-0085-4. PMID 11899300
- [Background] Newman DL, Hoffjan S, Bourgain C, Abney M, Nicolae RI, Profits ET, Grow MA, Walker K, Steiner L, Parry R, Reynolds R, McPeek MS, Cheng S, Ober C. Are common disease susceptibility alleles the same in outbred and founder populations? Eur J Hum Genet. 2004 Jul;12(7):584-90. doi: 10.1038/sj.ejhg.5201191. PMID 15100713
- [Background] Zollner S, Wen X, Hanchard NA, Herbert MA, Ober C, Pritchard JK. Evidence for extensive transmission distortion in the human genome. Am J Hum Genet. 2004 Jan;74(1):62-72. doi: 10.1086/381131. Epub 2003 Dec 15. PMID 14681832
- [Background] Weiss LA, Abney M, Cook EH Jr, Ober C. Sex-specific genetic architecture of whole blood serotonin levels. Am J Hum Genet. 2005 Jan;76(1):33-41. doi: 10.1086/426697. Epub 2004 Nov 3. PMID 15526234
- [Background] Kurz T, Ober C. The role of environmental tobacco smoke in genetic susceptibility to asthma. Curr Opin Allergy Clin Immunol. 2004 Oct;4(5):335-9. doi: 10.1097/00130832-200410000-00002. PMID 15349030
- [Background] McPeek MS, Wu X, Ober C. Best linear unbiased allele-frequency estimation in complex pedigrees. Biometrics. 2004 Jun;60(2):359-67. doi: 10.1111/j.0006-341X.2004.00180.x. PMID 15180661
- [Background] Hoffjan S, Nicolae D, Ober C. Association studies for asthma and atopic diseases: a comprehensive review of the literature. Respir Res. 2003 Dec 4;4(1):14. doi: 10.1186/1465-9921-4-14. Print 2003. PMID 14748924
- [Background] Nicolae D, Cox NJ, Lester LA, Schneider D, Tan Z, Billstrand C, Kuldanek S, Donfack J, Kogut P, Patel NM, Goodenbour J, Howard T, Wolf R, Koppelman GH, White SR, Parry R, Postma DS, Meyers D, Bleecker ER, Hunt JS, Solway J, Ober C. Fine mapping and positional candidate studies identify HLA-G as an asthma susceptibility gene on chromosome 6p21. Am J Hum Genet. 2005 Feb;76(2):349-57. doi: 10.1086/427763. Epub 2004 Dec 20. PMID 15611928
- [Background] Donfack J, Schneider DH, Tan Z, Kurz T, Dubchak I, Frazer KA, Ober C. Variation in conserved non-coding sequences on chromosome 5q and susceptibility to asthma and atopy. Respir Res. 2005 Dec 10;6(1):145. doi: 10.1186/1465-9921-6-145. PMID 16336695
- [Background] Ober C. HLA-G: an asthma gene on chromosome 6p. Immunol Allergy Clin North Am. 2005 Nov;25(4):669-79. doi: 10.1016/j.iac.2005.08.001. PMID 16257632
- [Background] Ober C, Thompson EE. Rethinking genetic models of asthma: the role of environmental modifiers. Curr Opin Immunol. 2005 Dec;17(6):670-8. doi: 10.1016/j.coi.2005.09.009. Epub 2005 Oct 7. PMID 16214315
- [Background] Ober C. Perspectives on the past decade of asthma genetics. J Allergy Clin Immunol. 2005 Aug;116(2):274-8. doi: 10.1016/j.jaci.2005.04.039. PMID 16083779
- [Background] Shilling RA, Pinto JM, Decker DC, Schneider DH, Bandukwala HS, Schneider JR, Camoretti-Mercado B, Ober C, Sperling AI. Cutting edge: polymorphisms in the ICOS promoter region are associated with allergic sensitization and Th2 cytokine production. J Immunol. 2005 Aug 15;175(4):2061-5. doi: 10.4049/jimmunol.175.4.2061. PMID 16081771
- [Background] Zhang J, Schneider D, Ober C, McPeek MS. Multilocus linkage disequilibrium mapping by the decay of haplotype sharing with samples of related individuals. Genet Epidemiol. 2005 Sep;29(2):128-40. doi: 10.1002/gepi.20081. PMID 16049966
- [Background] Kurina LM, Weiss LA, Graves SW, Parry R, Williams GH, Abney M, Ober C. Sex differences in the genetic basis of morning serum cortisol levels: genome-wide screen identifies two novel loci specific to women. J Clin Endocrinol Metab. 2005 Aug;90(8):4747-52. doi: 10.1210/jc.2005-0384. Epub 2005 Jun 7. PMID 15941864
- [Background] Weiss LA, Lester LA, Gern JE, Wolf RL, Parry R, Lemanske RF, Solway J, Ober C. Variation in ITGB3 is associated with asthma and sensitization to mold allergen in four populations. Am J Respir Crit Care Med. 2005 Jul 1;172(1):67-73. doi: 10.1164/rccm.200411-1555OC. Epub 2005 Apr 7. PMID 15817799